CLINICAL TRIAL: NCT01226212
Title: Can Synbiotic Use Improve Dysbiosis in the Gut Microbiome and Modify Inflammatory Processes in Older People
Brief Title: Can Synbiotic Use Effect Gut Bacteria and the Immune Response in Older People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: Chief Scientist Office of the Scottish Government (Other Government)
Responsible Party: Professor George Macfarlane, University of Dundee
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2010GA03; Funder (Other Grant/Funding Number: Chief Scientist Office ETM66)
Record Dates: First submitted 2010-10-18; First posted 2010-10-22 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-04

CONDITIONS: Aging
Keywords: Older people; Synbiotic; Prebiotic; Probiotic; Bacteria; Immune
MeSH Terms: interventions — Synbiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Synbiotic (Experimental): Synbiotic (Synergy 1/B. longum)
  Interventions: Dietary Supplement: Synbiotic (Synergy 1/B. longum)
- Placebo (Placebo Comparator): maltodextrose
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Synbiotic (Synergy 1/B. longum) — Combination of a prebiotic Synergy 1 and a probiotic Bifidobacterium longum
  Arms: Synbiotic
Dietary Supplement: Placebo — maltodextrose
  Arms: Placebo

SUMMARY:
The objectives of this study are to use a nutritional change in the diet to improve gut health in older people. Ageing can result in major changes in the composition and activities of the bacteria in your gut, leading to a higher incidence of gastrointestinal infections, decreased intestinal motility and impaired bowel function as people get older. This can result in constipation or diarrhoea, increased levels of inflammation and reduced immune response to infection. Therefore, individuals aged 65 or over could benefit from safe and effective interventions that maintain a healthy balance of gut bacteria as well as restoring the immune response. Bacteria in the gut are known to promote health. Eating foods containing beneficial bacteria for example (probiotics) or food which contain substrates for the bacteria to grow on (prebiotics) can improve the balance of gut bacteria. The investigators will use a synbiotic with known anti-inflammatory properties, comprising a probiotic Bifidobacterium longum strain and inulin (Synergy 1), The synbiotic has been previously shown to be beneficial in reducing inflammation and to increase levels of beneficial bacteria in the gut in two studies in patients with inflammatory bowel disease. The investigators would now for these reasons, like to determine the effects of our Synbiotic on the gut bacteria and immune function of older individuals in a double-blinded, crossover, placebo controlled, randomised investigation involving 40 volunteers for three months. The trial is designed so that participants will be assigned to receive the Synbiotic preparation or the placebo for the first four weeks, this will be followed by four weeks without treatment, and then they will switch to the opposite preparation for another four weeks.

ELIGIBILITY:
Inclusion Criteria:

* 65-90 years
* BMI 18.5-30.0 kg m2.

Exclusion Criteria:

* asplenia and other acquired or congenital immunodeficiencies
* any autoimmune disease
* connective tissue diseases
* self-reported symptoms of acute or recent infection (including use of antibiotics within the previous 3 months)
* taking probiotics or prebiotics, including lactulose for constipation
* chronic gastrointestinal problems (e.g. Inflammatory bowel disease, irritable bowel syndrome, cancer)
* use of immunosuppressive or anti-inflammatory drugs.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 49 (Actual)
Dates: Start 2010-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Increase in levels of faecal bifidobacteria | 4 weeks

SECONDARY OUTCOMES:
Improvement in inflammatory markers linked to ageing | 4 weeks
Improvement in bowel habit and quality of life | 4 weeks
Reduction of genotoxic potential | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: George Macfarlane, PhD, Principal Investigator — University of Dundee
Locations (1):
- Department of Oncology and Molecular Medicine, Ninewells Hospital and Medical School, Dundee, Tayside, United Kingdom

REFERENCES:
- [Background] Steed H, Macfarlane GT, Blackett KL, Bahrami B, Reynolds N, Walsh SV, Cummings JH, Macfarlane S. Clinical trial: the microbiological and immunological effects of synbiotic consumption - a randomized double-blind placebo-controlled study in active Crohn's disease. Aliment Pharmacol Ther. 2010 Oct;32(7):872-83. doi: 10.1111/j.1365-2036.2010.04417.x. PMID 20735782
- [Background] Macfarlane GT, Steed H, Macfarlane S. Bacterial metabolism and health-related effects of galacto-oligosaccharides and other prebiotics. J Appl Microbiol. 2008 Feb;104(2):305-44. doi: 10.1111/j.1365-2672.2007.03520.x. PMID 18215222
- [Background] Macfarlane S, Macfarlane GT, Cummings JH. Review article: prebiotics in the gastrointestinal tract. Aliment Pharmacol Ther. 2006 Sep 1;24(5):701-14. doi: 10.1111/j.1365-2036.2006.03042.x. PMID 16918875
- [Background] Furrie E, Macfarlane S, Kennedy A, Cummings JH, Walsh SV, O'neil DA, Macfarlane GT. Synbiotic therapy (Bifidobacterium longum/Synergy 1) initiates resolution of inflammation in patients with active ulcerative colitis: a randomised controlled pilot trial. Gut. 2005 Feb;54(2):242-9. doi: 10.1136/gut.2004.044834. PMID 15647189
- [Background] Woodmansey EJ, McMurdo ME, Macfarlane GT, Macfarlane S. Comparison of compositions and metabolic activities of fecal microbiotas in young adults and in antibiotic-treated and non-antibiotic-treated elderly subjects. Appl Environ Microbiol. 2004 Oct;70(10):6113-22. doi: 10.1128/AEM.70.10.6113-6122.2004. PMID 15466557
- [Background] Bartosch S, Fite A, Macfarlane GT, McMurdo ME. Characterization of bacterial communities in feces from healthy elderly volunteers and hospitalized elderly patients by using real-time PCR and effects of antibiotic treatment on the fecal microbiota. Appl Environ Microbiol. 2004 Jun;70(6):3575-81. doi: 10.1128/AEM.70.6.3575-3581.2004. PMID 15184159
- [Derived] Macfarlane S, Cleary S, Bahrami B, Reynolds N, Macfarlane GT. Synbiotic consumption changes the metabolism and composition of the gut microbiota in older people and modifies inflammatory processes: a randomised, double-blind, placebo-controlled crossover study. Aliment Pharmacol Ther. 2013 Oct;38(7):804-16. doi: 10.1111/apt.12453. Epub 2013 Aug 20. PMID 23957631